CLINICAL TRIAL: NCT03767179
Title: Research of Serum Procalcitonin, Erythrocyte Sedimentation Rate, C-Reactive Protein And Leukocyte Levels in Fertile Missed Abortion Cases
Brief Title: Research of Serum Procalcitonin, ESR, CRP And Leukocyte Levels in Fertile Missed Abortion Cases
Status: Completed | Type: Observational
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Suleyman Guven, Clinical Professor., Karadeniz Technical University
Other Study IDs: KTU
Record Dates: First submitted 2018-06-17; First posted 2018-12-06 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Abortion, Missed
Keywords: Missed abortion; Procalcitonin; Erythrocyte sedimentation rate (ESR); C-reactive protein (CRP); Leukocyte (WBC)
MeSH Terms: conditions — Abortion, Missed

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood Serum, abortion materials
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group: The study group consisted of 30 fertile, under 35 years old women who were included in the study for the first time missed abortus diagnosis.
  Interventions: Diagnostic Test: study
- Control Group: 30 cases with the same trimester, fertile, and under 35 years old who were referred to Obstetrics clinic, who had no systemic disease, were included in the study.
  Interventions: Diagnostic Test: study

INTERVENTIONS:
Diagnostic Test: study — procalcitonin, sedimentation, CRP, leukocyte identification

SUMMARY:
Aim: The serum procalcitonin, erythrocyte sedimentation rate, c-reactive protein and leukocyte values will be compared between fertile missed abortion diagnosed pregnants and fertile normal pregnants to determine the presence of subclinical infection in the etiology of missed abortion

DETAILED DESCRIPTION:
The study group will consist of 30 fertile, under 35 years old women having for the first time missed abortus diagnosis in the Obstetrics Department of Obstetrics and Gynecology of Medicine Faculty of Karadeniz Technical University, Medical Faculty of Medicine. As control group, 30 cases with the same trimester, fertile, and under 35 years old who had referred to Obstetrics clinic, who had no systemic disease, will be included in the study. Blood samples will be collected at the time of diagnosis of the patients with missed abortion and in normal pregnancy in the week of 20th gestational week and will send to Biochemistry laboratory to examine procalcitonin, erythrocyte sedimentation rate, c-reactive protein and leukocyte values in their sera. The age, weight, gestational week, gravida (number), parity (number), abortus (number), body mass index, systemic diseases, blood group, smoking information, binary test results, and results of genetic analysis will be collected in both groups. The pathology results of the missed abortion group will also be collected. The results will statistically be compared in the SPSS 13.0 program in both groups.

ELIGIBILITY:
Inclusion Criteria:

* fertile, less than 20 weeks of geese who have missed abortus for the first time without systemic disease

Exclusion Criteria:

* Failure to meet the missed abortus diagnostic criteria (for the group of fertile missed abortus)
* Smoking
* Rejection to participate in the study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 60 pregnant women
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-04-15 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
Serum LC | 01.01.2018- 15.02.2019
  Serum leukocyte count in number
CRP | 01.01.2018- 15.02.2019
  Serum CRP level in microgram
ESR | 01.01.2018- 15.02.2019
  Erythrocyte sedimentation rate
Prokalsitonin | 01.01.2018- 15.02.2019
  Serum procalcitonin level in microgram

CONTACTS AND LOCATIONS:
Overall Officials: Suleyman Guven, Prof, Principal Investigator — KaradenizTU Medicine Faculty
Locations (1):
- Karadeniz Technical University, Medical Faculty of Medicine., Trabzon, Ortahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No